CLINICAL TRIAL: NCT02805686
Title: " En Face " OCT's Contribution in the Detection of Macular Retinal Toxicity Signs Linked to the Chronic Treatment of Synthetic Antimalarials
Acronym: OCTAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MMT_2014-7
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Maculopathy
Keywords: Toxicity, Drug
MeSH Terms: conditions — Macular Degeneration; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "En face" OCT (C-scan) (Experimental)
  Interventions: Device: spectral domain optical coherence tomography; Device: multifocal electroretinogram

INTERVENTIONS:
Device: spectral domain optical coherence tomography
Device: multifocal electroretinogram

SUMMARY:
The maculopathy induced by the retinal toxicity of the synthetic antimalarials must be detected at the infra-clinical state, when it can still be reversible. Identifying early retinal anatomical changes has always represented (a challenge for medical interns, dermatologists, rheumatologists, and ophthalmologists). Currently, the gold-standard for its screening and its diagnostic is the multifocal electroretinogram (mfERG), however it is a long and tedious exam, offered by only few medical centers. It is recommended to find a simple non-invasive alternative, on a commonly used equipment. The study of the ellipsoid (junction line between, the external and internal photoreceptor segments) using optical coherence tomography (OCT-SD) "en face" enables us, to obtain a panoramic viewing of the state of the photoreceptor layer, and to detect any modification, even subtle, within this layer. The OCT-SD "en face" can be easily done by any ophthalmologist who owns one.

The proportion of "en face" OCT-SD showing suggestive retinal damage and patients who present retinal damage in relation with synthetic antimalarial treatments and diagnosed by mfERG is considered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with synthetic antimalarials with retinal damage (in relation with the antimalarial treatment) recently diagnosed by mfERG
* Patients treated with synthetic antimalarials in the past, who stopped treatment because of a supposed retinal damage not confirmed by mfERG

Exclusion Criteria:

- State of ocular structures preventing the realization of exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
concordance between mfERG and "En-face" OCT | after 1 hour
  measure of kappa coefficient